CLINICAL TRIAL: NCT03740178
Title: A Randomized, Double-Blinded Clinical Trial to Assess the Safety, Tolerability and Pharmacokinetics of MK-4334 in Participants With Alzheimer's Clinical Syndrome on a Stable Dose of Donepezil
Brief Title: Multiple Dose Trial of MK-4334 in Participants With Alzheimer's Clinical Syndrome (MK-4334-005)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Development program discontinuation
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4334-005; MK-4334-005 (Other: Merck Protocol Number)
Record Dates: First submitted 2018-11-12; First posted 2018-11-14 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Alzheimer's Disease; Mild Cognitive Impairment
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — Donepezil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Donepezil + MK-4334 (Experimental): Oral MK-4334 60/120 mg QD and open-label, oral donepezil 10 mg QD.
  Interventions: Drug: MK-4334; Drug: Donepepzil
- Donepezil + Placebo (Placebo Comparator): Placebo to MK-4334 QD and open-label, oral donepezil 10 mg QD.
  Interventions: Drug: Placebo to MK-4334; Drug: Donepepzil

INTERVENTIONS:
Drug: MK-4334 — Participants with Alzheimer's clinical syndrome (MCI or mild/moderate AD) will receive MK-4334 capsules administered orally, QD on Days 1-14. Participants will receive an initial loading dose of 120 mg (Day 1), followed by a maintenance dose of 60 mg (Days 2-14). Open-label donepezil tablets (dose strength: 10 mg) administered orally, QD on Days 1-14.
  Other Names: Aricept
  Arms: Donepezil + MK-4334
Drug: Placebo to MK-4334 — Participants with Alzheimer's clinical syndrome (MCI or mild/moderate AD)will receive placebo capsules matching MK-4334 administered orally, QD on Days 1-14. Participants will also receive open-label donepezil tablets (dose strength: 10 mg) administered orally, QD on Days 1-14.
  Other Names: Aricept
  Arms: Donepezil + Placebo
Drug: Donepepzil — Participants with Alzheimer's clinical syndrome (MCI or mild/moderate AD) will receive open-label, oral donepezil 10 mg QD on Days 1-14.
  Other Names: Aricept

SUMMARY:
This study will evaluate the safety, tolerability, and pharmacokinetics of MK-4334 administered once daily (QD) in participants with Alzheimer's clinical syndrome receiving a stable, daily dose of donepezil 10 mg, taken orally (PO). This includes participants with symptoms of mild cognitive impairment (MCI) or mild to moderate Alzheimer's disease (AD). It is hypothesized that the true geometric mean minimum plasma concentration at 24 hours (C24) is at least 60 nM at steady state in the presence of steady-state donepezil 10 mg.

ELIGIBILITY:
Inclusion Criteria:

Participants with MCI

* Have a history of subjective memory decline with gradual onset and slow progression for at least one year before screening.
* Have general cognitive function and activities of daily living sufficiently intact, based on clinical assessment, so as not to meet criteria for mild AD dementia based on National Institute of Neurological and Communicative Diseases and Stroke/Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria.
* Have a Mini Mental State Exam-2 (MMSE-2) score ≥24.
* Have a Clinical Dementia Rating (CDR) scale score of 0.5, including a memory subscale score ≥ 0.5.

Participants with AD

* Have a history of cognitive and functional decline with gradual onset and slow progression for at least one year before screening.
* Meet the criteria for a diagnosis of probable AD based on NINCDS-ADRDA criteria.
* Have a MMSE-2 score ≥ 12 to ≤ 24 at screening.
* Have a CDR score of 1 to 2.

All Participants

* Have a Rosen-Modified Hachinski score ≤ 4.
* Be on a stable dose of donepezil 10 mg PO daily for symptomatic treatment of Alzheimer's clinical syndrome. The dose must be stable for ≥2 months prior to screening.
* Be in good health based on medical history, physical examination, vital sign (VS) measurements and electrocardiograms (ECGs) performed prior to randomization.
* Have a Body Mass Index (BMI) ≤ 35 kg/m^2.
* If female, is a woman of non-childbearing potential (WONCBP).
* If male, must agree to either remain abstinent or use contraception during the intervention period and for ≥28 days after the last dose of study intervention.
* Have acceptable venous access.

Exclusion Criteria:

* Is at imminent risk of self-harm, based on clinical interview and responses on the Columbia-Suicide Severity Rating Scale (C-SSRS), or of harm to others in the opinion of the investigator.
* Has a history of uncontrolled endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological (including stroke and chronic seizures) abnormalities or diseases.
* Has evidence of a clinically relevant or unstable psychiatric disorder, based on Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) criteria, including schizophrenia or other psychotic disorder, bipolar disorder, or delirium, at the time of prestudy (screening) visit, or has a history of clinically significant psychiatric disorder of the last 5 years.
* Has a history of cancer (malignancy), except for: 1.) adequately-treated nonmelanomatous skin carcinoma or carcinoma in situ of the cervix or; 2.) Other malignancies which have been successfully treated with appropriate follow up and therefore unlikely to recur for the duration of the study.
* Participant has an estimated creatinine clearance (CrCl) ≤55 mL/min based on the Modification of Diet in Renal Disease (MDRD).
* Has a history of significant multiple and/or severe allergies (e.g., food, drug, latex allergy), or has had an anaphylactic reaction or significant intolerability (i.e., systemic allergic reaction) to prescription or non-prescription drugs or food.
* Is positive for hepatitis B surface antigen, hepatitis C antibodies or human immunodeficiency virus (HIV).
* Had major surgery, donated or lost 1 unit of blood (approximately 500 mL) within 4 weeks prior to the prestudy (screening) visit.
* Is unable to refrain from or anticipates the use of strong or moderate inhibitors or inducers of Cytochrome P450 (CYP) 3A4 (CYP3A4) and CYP2C19 beginning approximately 28 days prior to administration of the initial dose of study drug, throughout the study, and until the post-trial visit.
* Has participated in another investigational study within 4 weeks (or 5 half-lives, whichever is greater) prior to the prestudy (screening) visit.
* Has a rate-corrected QT (QTc) interval ≥470 msec (for males) or ≥480 msec (for females).
* Is a smoker and/or has used nicotine or nicotine-containing products (e.g., nicotine patch and electronic cigarette) within 3 months of screening.
* Consumes greater than 3 glasses of alcoholic beverages (1 glass is approximately equivalent to: beer [354 mL/12 ounces], wine [118 mL/4 ounces], or distilled spirits [29.5 mL/1 ounce]) per day.
* Consumes excessive amounts, defined as greater than 6 servings of coffee, tea, cola, energy drinks, or other caffeinated beverages per day.
* Is a regular user of cannabis, any illicit drugs or has a history of drug (including alcohol) abuse within approximately 2 years. Participants must have a negative urine drug screen prior to randomization.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09-27 (Estimated); Primary Completion 2020-02-28 (Estimated); Study Completion 2020-02-28 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Experiencing an Adverse Event (AE) | Up to 42 days
  An AE is any unfavorable and unintended sign, symptom, or disease (new or exacerbated) in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study treatment. For each arm, the number of participants experiencing an AE will be assessed.
Number of Participants Discontinuing Study Treatment due to an Adverse Event | Up to 14 days
  An AE is any unfavorable and unintended sign, symptom, or disease (new or exacerbated) in a clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. For each arm, the number of participants discontinuing study treatment due to an AE will be assessed.

SECONDARY OUTCOMES:
Plasma Steady State Concentration at 24 Hours (C24) of MK-4334 | Day 14: Pre-dose and 24 hours after MK-4334 administration
  Plasma steady state concentration at 24 hours (C24) will be reported.
Plasma Steady State Area Under the Concentration-Time Curve from 0 to 24 hours (AUC0-24) of MK-4334 | Day 14: Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, and 24 hours after MK-4334 administration
  Plasma steady state area under the concentration-time curve from 0 to 24 hours (AUC0-24) will be reported.
Plasma Steady State Maximum Concentration (Cmax) of MK-4334 | Day 14: Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 120, 240, 360, and 480 hours after MK-4334 administration
  Plasma steady state maximum concentration (Cmax) will be reported.
Plasma Steady State Apparent Half-Life (t1/2) of MK-4334 | Day 14: Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 120, 240, 360, and 480 hours after MK-4334 administration
  Plasma steady state apparent half-life (t1/2) will be reported.
Plasma Steady State Time to Maximum Concentration (Tmax) of MK-4334 | Day 14: Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 120, 240, 360, and 480 hours after MK-4334 administration
  Plasma steady state time to maximum concentration (Tmax) will be reported.
Plasma Steady State Apparent Clearance (CL/F) of MK-4334 | Day 14: Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 120, 240, 360, and 480 hours after MK-4334 administration
  Plasma steady state apparent clearance (CL/F) will be reported.
Plasma Steady State Apparent Volume of Distribution (Vz/F) of MK-4334 | Day 14: Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 120, 240, 360, and 480 hours after MK-4334 administration
  Plasma steady state apparent volume of distribution (Vz/F) will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/